CLINICAL TRIAL: NCT05378841
Title: Efficacy of Surgical Joint Denervation in Painful Digital Osteoarthritis
Acronym: DECAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP211437; 2022-A00794-39 (Other: IDRCB)
Record Dates: First submitted 2022-04-15; First posted 2022-05-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis Hand
Keywords: Digital osteoarthritis; Surgical joint dernervation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical denervation (Experimental): It consists of a section of the nerve branches destined for the PIPJ, coming from the digital collateral nerves as well as the dorsal sensory branches of the radial and ulnar nerves respectively for the index and fifth fingers.
  Interventions: Procedure: Surgical Denervation

INTERVENTIONS:
Procedure: Surgical Denervation — This is an outpatient procedure performed under local anesthesia (depending on the anesthesiologist's decision), which lasts about 30 minutes.

SUMMARY:
Digital osteoarthritis is the second localization of symptomatic osteoarthritis, after the knee. Its cardinal symptoms are particularly intense pain and functional impairment in the case of the erosive form. There is currently no etiological treatment for osteoarthritis. Symptomatic treatments have a modest efficacy, which justifies the search for new treatments. The surgical options are arthrodesis or prosthesis, invasive techniques potentially sources of complications, and finally proposed infrequently given the prevalence of digital osteoarthritis.

DECAD is a prospective phase II trial aimed at evaluating the efficacy of surgical joint denervation in painful digital osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is the most common joint pathology of the musculoskeletal system. It affects 6 million French people and constitutes a public health problem. Osteoarthritis of the hands or digitalis is the second localization of symptomatic osteoarthritis, after the knee. Its main risk factors are female sex, age, genetic factors, and obesity.

Osteoarthritis combines articular cartilage degradation, synovial inflammation, subchondral bone remodeling and osteophyte development. Its cardinal symptoms are pain and functional impairment (at a level sometimes close to inflammatory rheumatism such as rheumatoid arthritis), particularly intense in the case of the erosive form. There is also local joint inflammation associated with pain. Pain in osteoarthritis is a complex phenomenon involving joint tissues other than cartilage, a tissue that is not innervated (subchondral bone, joint capsule, synovial membrane).

There is currently no etiological treatment for osteoarthritis. Symptomatic treatments have a modest efficacy, which justifies the search for new treatments. The surgical options are arthrodesis or prosthesis, invasive techniques potentially sources of complications, and finally proposed infrequently given the prevalence of digital osteoarthritis.

The only current conservative surgical solution that can be proposed for intractable painful proximal interphalangeal joint (PIPJ) osteoarthritis is denervation. This technique consists of cutting the nerve branches intended for the PIPJ in order to directly interrupt the pain pathways. It reduces pain by 80% after 5 years, without loss of mobility. There are only 4 published series reporting the results of this technique (2-3). These were retrospective case series with a low level of evidence. The patient satisfaction rate reached 90%, with transient paresthesias as the only reported complication. The mechanism of action for the effectiveness of this intervention has never been studied.

Our hypothesis is that denervation of the PIP has clinical efficacy in painful digital osteoarthritis refractory to usual treatments, and that it would have a structural effect that can be objectified on MRI.

The results of this pilot study will make it possible to construct a prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with symptomatic digital osteoarthritis according to the criteria of the American College of Rheumatology
* 1 painful PIP joint (Analog digital scale ≥ 4/10) for more than 3 months
* having failed the usual medical treatment for a minimum of 3 months (level 1 analgesics, NSAIDs, infiltrations)
* Signature of informed consent
* patient affiliated to a social security scheme
* knowing how to read French (for the questionnaires)

Exclusion Criteria:

* digital osteoarthritis secondary to other known causes (eg gout, reactive arthritis, RA, psoriatic arthritis, spondyloarthropathies, septic arthritis)
* anesthetic contraindications to surgery or to performing an MRI
* Existence of a pain syndrome in the upper limbs, which would interfere with the assessment of AD.
* Fibromyalgia
* Use of oral, intramuscular or intra-articular or intravenous corticosteroids, immunosuppressants (methotrexate, sulfasalazine, leflunomide, biomedicines), hyaluronic acid infiltration in the finger joints in the previous month
* Introduction of a new treatment for osteoarthritis of the hand in the previous month, including physiotherapy and fitting of a new finger orthosis.
* History of denervation of the proximal interphalangeal joint (PIP)
* Patient under legal protection (guardianship or curatorship) and patient deprived of liberty
* Patient under AME
* Participation in another interventional research involving the human person or period of exclusion at the end of a previous research involving the human person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Success of the intervention at 3 months | 3 months
  Success of the intervention at 3 months, defined by a reduction in pain of at least 2 points compared to the measurement at inclusion, with the numerical painscale (from 0 to 10) for the operate finger

SECONDARY OUTCOMES:
Pain at 6 months | 6 months
  Assessement with Numerical pain scale of the operated finger and the operated hand (from 0 to 10)
Quality of life at 6 months : Score quick-DASH | 6 months
  Calculation of score by quick-DASH questionnary: main functional and quality of life and function score used in hand surgery
Quality of life at 6 months : Score AUSCAN | 6 months
  Calculation of score by AUSCAN questionnary (Australian/Canadian Osteo Arthritis Hand Index, self-administered questionnaire validated in AD measuring pain, function and stiffness)
Grip strength at 6 months | 6 months
  Grip strength measured by JAMAR hydraulic dynamometer to assess the impact of pain on function
PGI-C Score at 6 months | 6 months
  Calculation of score on PGI-C scale (Patient Global Impressions scale-Change, assesses the perception of a change induced by the treatment) to assess patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie SELLAM, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Rheumatology department Saint-Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided